CLINICAL TRIAL: NCT06975969
Title: Single Center Post-Market Study of Thrombolytic Therapy Using the Versus™ Catheter
Status: Recruiting | Type: Observational
Sponsor: Liquet Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1001; 1402 Liquet-UVA-VCU (Other Grant/Funding Number: VBHRC Catalyst)
Record Dates: First submitted 2025-04-23; First posted 2025-05-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Blood Clots; Vascular Disease; Embolism Thrombosis; Cardiovascular Diseases; Lung Diseases
Keywords: thrombolysis; pulmonary catheter; hemodynamic monitoring; catheter directed therapy
MeSH Terms: conditions — Thrombosis; Vascular Diseases; Embolism and Thrombosis; Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who receive treatment using the Versus Catheter: Patients age 18 - 80 years old who present with symptoms requiring intervention with delivery of physician-specified thrombolytics to the pulmonary vasculature, including patients who present with submassive pulmonary embolism (PE), who receive treatment using the Versus™ Catheter.
  Interventions: Device: Versus™ Endovascular Pulmonary Artery Drug Delivery Catheter

INTERVENTIONS:
Device: Versus™ Endovascular Pulmonary Artery Drug Delivery Catheter — The Versus Pulmonary Artery Catheter is a dual-tip, infusion catheter. Two lumens access and deliver physician-specified fluids, including thrombolytics, into the pulmonary arteries of each lung via a single access site. The Secondary Catheter tip telescopes independently to facilitate infusion into the contralateral lung. The device may allow for assessment of a patient's hemodynamic condition through direct intracardiac and pulmonary artery pressure monitoring. Pressure is measured through an interface between the catheter's fluid lumen and an externally located, FDA-cleared, pressure transducer. The device may include an additional lumen that is in communication with a distal flow-directed balloon.

SUMMARY:
Assess the functionality of the Versus Catheter for catheter-directed thrombolysis of pulmonary blood clots, including advanced imaging assessment. An evaluation of patient outcomes from the cases included in this study will also be conducted.

DETAILED DESCRIPTION:
The objective of this study is to assess the functionality of the Versus™ Catheter for the controlled and selective infusion of physician-specified fluids, including thrombolytics, into the pulmonary artery vasculature in adult patients, including advanced Computerized Tomography Angiogram (CTA) imaging assessment. This study will include an evaluation of patient outcomes and physician user experience with the Versus™ Catheter among up to 10 patients meeting the criteria for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 80 years, inclusive
* Patients who present with submassive pulmonary embolism (PE)
* Patients requiring thrombolytic intervention to the pulmonary vasculature
* Physician decision to use the Versus™ Catheter during the treatment of the patient

Exclusion Criteria:

* Concurrent treatment with thrombectomy
* Concurrent treatment with a catheter-directed thrombolysis device that is NOT the Versus™ Catheter
* Massive pulmonary embolism (PE)
* Active bleeding disorder1
* Recent cerebrovascular accident or transient ischemic attack1
* Recent neurosurgery1
* Recent intracranial trauma1
* Absolute contraindication to anticoagulation1
* BMI > 45kg/m2
* In the opinion of the investigator, the participant is not a suitable candidate for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 - 80 years old who present with symptoms requiring intervention with delivery of physician-specified thrombolytics to the pulmonary vasculature, including patients who present with submassive pulmonary embolism (PE), who receive treatment using the Versus™ Catheter.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Clot resolution | Within one week of hospital admission
  Number of patients achieving hemodynamic homeostasis as evidenced by pulmonary artery pressure indicating resolution of a pulmonary blood clot
Physician user experience | Periprocedural
  Number of physicians who rate use of the Versus Catheter as "Good & Acceptable" or "Very good & Acceptable" on a four-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Luke Wilkins, MD, Principal Investigator — University of Virgina (UVA)
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No